CLINICAL TRIAL: NCT01960816
Title: Pilot Study of Aerin Medical's InFlux System for Improvement in Nasal Breathing
Brief Title: InFlux System for Nasal Breathing Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP026
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-08

CONDITIONS: Nasal Airway Obstruction
Keywords: nasal obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- InFlux System (Experimental): Intervention: Procedure: thermal coagulation of tissue in the nasal airway
  Interventions: Device: Procedure: thermal coagulation of tissue in the nasal airway

INTERVENTIONS:
Device: Procedure: thermal coagulation of tissue in the nasal airway — The Vivaer Stylus is used to deliver low-power, temperature-controlled, radiofrequency energy to tissues of the nasal airway to cause coagulation of soft tissues and submucosal tissue shrinkage.
  Other Names: Vivaer Stylus; Aerin Medical Wand

SUMMARY:
Pilot Study of the Aerin Medical Wand used for Improvement in Nasal Breathing

DETAILED DESCRIPTION:
This is a non-significant risk, prospective, non-randomized pilot study to evaluate the incidence of serious adverse events directly attributable to the Aerin Medical Wand, when used to deliver radiofrequency (RF) energy to tissues of the nasal airway for the treatment of nasal obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of Chronic nasal obstruction and Poor nasal breathing

Exclusion Criteria:

* Patients with prior nasal history, nasal pathology, or injury, and/or other conditions that may interfere with participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Catalano, MD, Principal Investigator — Steward Hospital
Locations (2):
- United States (2):
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Bay Area ENT, Ocean Springs, Mississippi

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | InFlux System
Started | 33
Completed | 32
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | InFlux System
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 33
Nasal Obstruction Symptom Evaluation (NOSE) score [Mean (Standard Deviation); unit: units on a scale] — The Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific health status outcomes instrument, used to assess severity of nasal obstruction symptoms. Score ranges from 0 to 100. Higher scores indicate increased symptoms/symptom severity.
  units on a scale | 58 (21.8)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Unanticipated Serious Adverse Device Effects
Description: The study will be considered to have met its primary safety endpoint if no subject experiences an unanticipated serious adverse device effect (USADE defined as any serious adverse effect caused by, or associated with, the investigational device, that was not previously identified in nature, severity, or degree of incidence in the protocol)
Time Frame: 90 Days
Population: One subject was lost-to-follow-up prior to the 90-day follow-up visit. Therefore, 32 subjects were available for analysis at the 90-day time point.
Measure: Number; unit: events
Arm/Group | InFlux System
Number analyzed (Participants) | 32
events | 0

2. Primary Outcome: Technical Feasibility as Assessed by the Ability of the InFlux Device to Deliver RF Energy to Target Tissue
Description: Ability of the InFlux device to deliver RF energy at the selected power setting, and to reach and maintain the selected target temperature.
Time Frame: Procedure, up to 1 hour (average, 16 minutes)
Population: All enrolled subjects underwent the procedure.
Measure: Number; unit: participants
Arm/Group | InFlux System
Number analyzed (Participants) | 33
participants | 33

3. Post Hoc Outcome: NOSE Score at 90-day Follow-up
Description: The Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific health status outcomes instrument, used to assess severity of nasal obstruction symptoms. Score ranges from 0 to 100. Higher scores indicate increased symptoms/symptom severity. Each subject's NOSE score at the 90-day follow-up was compared to that subject's baseline NOSE score to determine change in nasal obstruction symptoms.
Time Frame: 90 days
Population: Subjects with 90-day follow-up data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | InFlux System
Number analyzed (Participants) | 32
units on a scale | 27 (21.1)

ADVERSE EVENTS:
Arm/Group | InFlux System
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 2/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InFlux System (N=33)
Upper respiratory infection / symptoms of common cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Adverse events deemed not related to the investigational device or procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less